CLINICAL TRIAL: NCT02027038
Title: Pelvic Belt Effects on Osseous Anatomy, Muscule Activation and Ground Reaction Forces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Bauerfeind AG, Zeulenroda-Triebes (Unknown)
Responsible Party: Principal Investigator, Niels Hammer, Dr. Niels Hammer, M.D., University of Leipzig
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 063/11/07032011
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Sacroiliac Joint Pain; Helath Related Quality of Life; Electromuscular Activation of the Pelis and Limbs; Ground Reaction Force Data

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with sacroiliac joint pain (Experimental): Patients suffering from sacroiliac joint pain
  Interventions: Device: Pelvic belt application
- Controls (Active Comparator): healthy controls
  Interventions: Device: Pelvic belt application

INTERVENTIONS:
Device: Pelvic belt application

SUMMARY:
Hypothesis I: The anatomic alignment of the pelvic bones, the electromuscular activation of limb muscles and ground reaction forces are different in patients with sacroiliac joint pain, as compared to healthy controls.

Hypothesis II: The application of pelvic belts alters the alignment of the pelvic bones, the electromuscular activation of the limb muscles or ground reaction forces.

Hypothesis III: The effects proposed in hypothesis II are different in patients with sacroiliac joint pain, as compared to healthy controls.

DETAILED DESCRIPTION:
The sacroiliac joint is among the most frequently involved anatomical structure in low back pain. Pelvic belt anatomy makes the sacroiliac joint more vulnerable to be involved in chronic painful conditions. However, the anatomical and functional correlate of sacroiliac joint pain is yet undetermined. According to the guidelines of International Association for the Study of Pain (IASP), painful conditions should primarily be managed conservatively.

However, existing studies fail providing sound evidence on the effects of conservative devices to therapy sacroiliac joint pain. In the study, a total of 17 patients suffering from sacroiliac joint pain and 17 controls were investigated by means of magnetic resonance imaging, EMG, health surveys and ground reaction force measurements.

A pelvic compression belt was administered in two levels of compression and the corresponding magnetic resonance imaging, EMG and ground reaction force data were measured.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnostically confirmed sacroiliac joint pain
* controls without any history of musculoskeletal disorders

Exclusion Criteria:

* endoprostheses, metallic implants
* somatoform disorders, claustrophobia, pregnancy
* surgical interventions on the spine, degenerative joint diseases elsewhere

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in pelvic bone alignment by pelvic belt, electromuscular activation, ground reaction force and in health outcome | 3-5 hours
  First application of pelvic belt = starting point No compression, moderate and maximum compression Health survey completion = end point

SECONDARY OUTCOMES:
Health related quality of life due to pelvic belt application | 6 weeks
  starting point: end of primary outcome measure ending point: 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Niels Hammer, M.D., Principal Investigator — University of Leipzig

REFERENCES:
- [Derived] Hammer N, Mobius R, Schleifenbaum S, Hammer KH, Klima S, Lange JS, Soisson O, Winkler D, Milani TL. Pelvic Belt Effects on Health Outcomes and Functional Parameters of Patients with Sacroiliac Joint Pain. PLoS One. 2015 Aug 25;10(8):e0136375. doi: 10.1371/journal.pone.0136375. eCollection 2015. PMID 26305790